CLINICAL TRIAL: NCT04653753
Title: Assessment of the Safety and Performance of a Patellofemoral Brace
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: kneeSOFT500
Record Dates: First submitted 2020-09-04; First posted 2020-12-04 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Patellofemoral Pain Syndrome; Patellar Instability
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthosis Group (Experimental): Use of kneeSOFT500 device
  Interventions: Device: kneeSOFT500
- Control Group (No Intervention): No use of the device

INTERVENTIONS:
Device: kneeSOFT500 — At least 30 patients (15 patients in the orthosis group and 15 patients in the control group) will be included. Patients included in the orthosis group will use the device during sports sessions while patients included in the control group will not use a knee support device.
  Arms: Orthosis Group

SUMMARY:
Decathlon has developed kneeSOFT500 product, which is a medical device intended to be used on the knee to keep a physical activity on a regular basis in case of patellofemoral pain syndrome or patellar instability. The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon kneeSOFT500 product to demonstrate safety and performance of this device in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥18 years old
* Subject has patellofemoral syndrome
* The current condition of his/her knee allows the subject to keep a regular physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (18 weeks)
* Subject is affiliated to the French social security regime

Non-Inclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (knee brace or articulated orthosis) in the last month during his/her sport practice
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (polyamide, cotton, elastane, elastodiene, polyester)
* Adult subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Functional score | 18 weeks of follow-up
  Comparison of the functional result (Kujala Anterior Knee Pain Scale, 0-100 points) between the baseline and last follow-up visit in each group (orthosis vs control)

SECONDARY OUTCOMES:
Confidence level | At baseline and 18 weeks of follow-up
  Gap in the confidence level (patient rated outcome with 6 questions, ranging from 0 to 100) related to physical activity, between the baseline and last follow-up visit in each group (orthosis vs control)
Knee instability | At 6 weeks, 12 weeks and 18 weeks of follow-up
  Comparison of knee instability, assessed through a numerical rating scale (NRS, ranging from 0 to 10), between the groups (orthosis vs control)
Knee pain | At 6 weeks, 12 weeks and 18 weeks of follow-up
  Comparison of knee pain, assessed through NRS (ranging from 0 to 10), between the groups (orthosis vs control)
Safety (adverse events) | 18 weeks of follow-up
  Comparison of adverse events rates between the groups (orthosis vs control)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (4):
- France (4):
  - Centre de rééducation et de balnéothérapie Kinés Faches, Faches-Thumesnil
  - Physio Sport Levallois, Levallois-Perret
  - Centre Hospitalier Universitaire de Lille, Lille
  - Cabinet de kinésithérapie du Belvédère, Paris

IPD SHARING:
Plan to Share IPD: No